CLINICAL TRIAL: NCT06421051
Title: Transauricular Vagus Nerve Stimulation (taVNS) Improves Postoperative Sleep Disorders in Elderly Patients:a Randomized Controlled Study.
Brief Title: Transauricular Vagus Nerve Stimulation Improves Postoperative Sleep Disorders in Elderly Patients.
Acronym: Vnstep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HX-B-2024016
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-07

CONDITIONS: Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high-frequency vagus nerve electrical stimulation (Experimental)
  Interventions: Device: Transauricular Vagal Nerve Stimulation
- low-frequency vagus nerve electrical stimulation (Placebo Comparator)
  Interventions: Device: Transauricular Vagal Nerve Stimulation

INTERVENTIONS:
Device: Transauricular Vagal Nerve Stimulation — Transauricular vagal nerve stimulation

SUMMARY:
Postoperative sleep disorder is one of the common complications after general anesthesia. Compared to patients of various ages, elderly patients have a much higher incidence of postoperative sleep disturbance. Postoperative sleep disorders can have many adverse effects, including cognitive impairment, altered pain perception, and emotional disorders, which are not conducive to the long-term prognosis of elderly patients. Enhancing postoperative sleep quality in older patients has become a significant public health concern in the current day due to its direct relationship to both maximizing surgical outcomes and enhancing physical health. This study intends to conduct a prospective, randomized controlled, triple-blind clinical trial on use of transauricular vagal nerve stimulation to improve sleep disorders in elderly patients after general anesthesia surgery, aiming to investigate the efficacy of transauricular vagal nerve stimulation in postoperative sleep disorders in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-craniocerebral surgery under elective general anesthesia
* Age ≥65 years old
* American society of Aneshesiologists Grade I to III
* Sign informed consent

Exclusion Criteria:

* Patients who are expected to retain tracheal intubation after surgery
* Disturbance of consciousness, mental disorder, inability to cooperate
* Expected survival < 3 months
* The estimated operation time is < 2 hours
* The expected postoperative hospital stay is < 5 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of sleep disorders within 5 days after surgery. | Day 1 to day 5 after surgery.

SECONDARY OUTCOMES:
Sleep quality after surgery. | Day 1,3,5 after surgery.
  The investigators collected patient-related information on postoperative days 1, 3, and 5 by using the Pittsburgh Sleep Quality Index (total score ranges from 0 to 21, with higher scores indicating poorer sleep quality) and a sleep monitoring bracelet, and analyzed the subsequent data.
Postoperative pain score | Day1 and 2 after surgery.
  The investigators collected information from the patients on the 1st and 2nd postoperative days by Visual Analogue Scale and analyzed the data subsequently. The scale is based on a 10-cm horizontal line drawn on a piece of paper, with 0 cm at one end of the line indicating "no pain at all" and 10 cm at the other end indicating "extreme pain"; the level of pain increases from 0 to 10 cm, with higher scores indicating more intense pain. The higher the score, the more severe the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang T, Wu Y, Hou X, Liang F, Jian M, Yu Y, Wang Y, Liu H, Han R. Transauricular vagus nerve electrical stimulation improves postoperative sleep disorders in elderly patients (VNstep): protocol for a randomized controlled clinical trial. Trials. 2026 Jan 21. doi: 10.1186/s13063-026-09459-z. Online ahead of print. PMID 41566492